CLINICAL TRIAL: NCT04191707
Title: Metabolomic Markers of Fatigue in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Diana Horta-Sangenis, principal investigator, Corporacion Parc Tauli
Other Study IDs: 2014068
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Fatigue; Inflammatory Bowel Disease; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Fatigue; Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 5 ml of peripheral blood by venepuncture into EDTA-K3 tubes (BD Biosciences, Spain). Plasma was separated by centrifugation of the samples at 2400 g for 10 min at 4°C and stored at - 80°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatients with Inflammatory Bowel Disease: This study was performed with plasma samples from IBD patients recruited in a previous study after informed consent. (1) IBD outpatients attending the Hospital de Sabadell Gastroenterology Day-care unit were consecutively included for analytical monitoring of immunosuppressant treatment or infliximab infusion

SUMMARY:
Fatigue is a common symptom and a leading concern in patients with inflammatory bowel disease (IBD) and often persists despite clinical and endoscopic remission.

This study evaluates the metabolomic profile of fatigued patients with IBD.

DETAILED DESCRIPTION:
To date, there is only one non-published study using metabolomics in quiescent IBD patients with and without fatigue.

The investogators designed this study to examine if there are metabolomics factors associated to fatigue in IBD patients.

This study was performed with plasma samples from IBD patients recruited in a previous study after informed consent. (1) IBD outpatients attending the Hospital de Sabadell Gastroenterology Day-care unit were consecutively included for analytical monitoring of immunosuppressant treatment or infliximab infusion.

The investigators recorded demographic data, IBD classification according to the Montreal classification, and history of drug administration. In addition, clinical activity of the disease was measured using the Harvey-Bradshaw score for Crohn's disease (CD) and the modified Mayo score for ulcerative colitis (UC). The "Functional Assessment of chronic Illness Therapy-Fatigue" (FACIT-F) was used to assess fatigue.

ELIGIBILITY:
Inclusion Criteria:

- Inflammatory bowel disease diagnosed at least 6 months before the study (diagnosed by clinical, laboratory , endoscopic and histological criteria) .

Exclusion Criteria:

* Age below 18 years.
* Refusal to give written informed consent prior to participation
* Active infection at the time of inclusion.
* Concomitant diseases not related to IBD (e.g., cancer, heart disease, pulmonary disease) that might contribute to the presence or the severity of fatigue.
* Active flare of IBD in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was performed with plasma samples from IBD patients recruited in a previous study after informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
changes in metabolomic profile | 1 year
  The metabolic profile consisted in 75 metabolites that were measured

CONTACTS AND LOCATIONS:
Overall Officials: Diana Horta, Principal Investigator — Parc Tauli Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villoria A, Garcia V, Dosal A, Moreno L, Montserrat A, Figuerola A, Horta D, Calvet X, Ramirez-Lazaro MJ. Fatigue in out-patients with inflammatory bowel disease: Prevalence and predictive factors. PLoS One. 2017 Jul 27;12(7):e0181435. doi: 10.1371/journal.pone.0181435. eCollection 2017. PMID 28749985